CLINICAL TRIAL: NCT01696435
Title: VITAL-DEP: Depression Endpoint Prevention in the VITamin D and OmegA-3 TriaL
Acronym: VITAL-DEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Olivia Okereke, Olivia I. Okereke, MD, SM, Principal Investigator, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-P-001881; R01MH091448 (NIH); R56MH091448 (NIH)
Record Dates: First submitted 2012-09-24; First posted 2012-10-01 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Depression; Depressive Symptoms; Mood
Keywords: Depression; Depressive Symptoms; Mood; Geriatric; Prevention
MeSH Terms: conditions — Depression | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil placebo (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator): Vitamin D placebo
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D placebo
- Vitamin D placebo + fish oil placebo (Active Comparator): Vitamin D placebo
  Fish oil placebo
  Interventions: Dietary Supplement: Fish oil placebo; Dietary Supplement: Vitamin D placebo
- Vitamin D + fish oil (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Dietary Supplement: vitamin D3; Drug: omega-3 fatty acids (fish oil)

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Other Names: fish oil
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Dietary Supplement: Vitamin D placebo — Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or fish oil: 1) reduces risk of clinical depressive syndrome, 2) yields better mood scores over time, compared to placebo.

DETAILED DESCRIPTION:
VITAL-DEP: Depression Endpoint Prevention in the VITamin D and OmegA-3 TriaL is a randomized clinical trial of vitamin D (in the form of vitamin D3 [cholecalciferol]) and marine omega-3 fatty acid (eicosapentaenoic acid [EPA] + docosahexaenoic acid [DHA]) supplements in the prevention of depression in older adults. Existing data from laboratory studies, epidemiologic research, limited clinical trials research suggest that these nutritional agents may reduce risk of depression or improve mood, but large primary prevention trials with adequate dosing and lengthy treatment durations in general populations are lacking.

Eligible participants will be assigned by chance (like a coin toss) to one of four groups: (1) daily vitamin D3 and omega-3; (2) daily vitamin D3 and omega-3 placebo; (3) daily vitamin D placebo and omega-3; or (4) daily vitamin D placebo and omega-3 placebo. Participants have an equal chance of being assigned to any of these four groups and a 3 out of 4 chance of getting at least one active agent.

Participants in all groups will take two pills each day -- one softgel that contains either vitamin D3 or vitamin D placebo and one capsule that contains either omega-3 or omega-3 placebo. Participants will receive their study pills in convenient calendar packages via U.S. mail.

Participants will also fill out a short (15-20 minute) questionnaire each year. The questionnaire asks about health; lifestyle habits such as physical exercise, diet, and smoking; use of medications and dietary supplements; family history of illness, and new medical diagnoses. The questionnaire also includes specific questions pertaining to mood. Occasionally, participants may receive a phone call from study staff to collect information or to clarify responses on the questionnaire.

Primary aims of 1) reduction in risk of clinical depressive syndrome and 2) yielding of better mood scores over time will be address in the full VITAL cohort of 20,000. Secondary aims will be addressed in sub-set of participants. The secondary aims will address whether: 1) among a subset of 1,000 participants evaluated at a Clinical and Translational Science Center (CTSC), the agents reduce risk of depression and yield better mood scores among persons with known risk factors for late-life depression; 2) among a subset of 1,000 participants evaluated at a CTSC, the agents reduce risk of major depression and yield better mood scores among persons with sub-syndromal depressive symptoms; 3) among all VITAL participants, African-American race (African-Americans have high risk of Vitamin D deficiency) modifies effects of vitamin D3 supplementation on late-life depression risk and on mood scores; 4) among a subset of participants, baseline plasma levels of vitamin D and omega-3 fatty acids are related to depression risk and/or modify agent effects.

Thus, VITAL-DEP will address simultaneously the impact of both vitamin D and fish oil for universal, selective and indicated prevention of late-life depression.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) who meet the following criteria are eligible to participate in this ancillary study. These are the criteria specific for testing of the primary aims in the VITAL-DEP ancillary study:

* no current significant depressive symptoms
* no core major depressive disorder symptoms for a period of two or more weeks in the past two years
* no history of alcohol and/or substance abuse disorder active in the past 12 months, schizophrenia or other primary psychotic disorder, bipolar disorder, post-traumatic stress disorder or obsessive-compulsive disorder
* no current psychotherapy or current use of psychotropics (including non-prescription agents for the treatment of mood disorders), except for limited use of mild sedatives/hypnotics
* no history of major neurologic disorder or delirium episode in the past 12 months
* no history of clinical (i.e., overt and not sub-clinical) hypothyroidism diagnosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18353 (Actual)
Dates: Start 2010-07; Primary Completion 2021-12-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia I Okereke, MD, SM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vyas CM, Kang JH, Mischoulon D, Cook NR, Reynolds Iii CF, Chang G, Mora S, De Vivo I, Manson JE, Okereke OI. Apolipoprotein E and Its Association With Cognitive Change and Modification of Treatment Effects of Vitamin D3 and Omega-3s on Cognitive Change: Results From the In-Clinic Subset of a Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2024 Mar 1;79(3):glad260. doi: 10.1093/gerona/glad260. PMID 37952113
- [Derived] Vyas CM, Mischoulon D, Chang G, Cook NR, Weinberg A, Copeland T, Kang JH, Bubes V, Friedenberg G, LeBoff MS, Lee IM, Buring JE, Manson JE, Reynolds CF, Okereke OI. Effects of Vitamin D3 and Marine Omega-3 Fatty Acids Supplementation on Indicated and Selective Prevention of Depression in Older Adults: Results From the Clinical Center Sub-Cohort of the VITamin D and OmegA-3 TriaL (VITAL). J Clin Psychiatry. 2023 Jun 26;84(4):22m14629. doi: 10.4088/JCP.22m14629. PMID 37378490
- [Derived] Vyas CM, Mischoulon D, Chang G, Reynolds CF 3rd, Cook NR, Weinberg A, Copeland T, Bubes V, Bradwin G, Lee IM, Buring JE, Mora S, Rifai N, Manson JE, Okereke OI. Relation of serum BDNF to major depression and exploration of mechanistic roles of serum BDNF in a study of vitamin D3 and omega-3 supplements for late-life depression prevention. J Psychiatr Res. 2023 Jul;163:357-364. doi: 10.1016/j.jpsychires.2023.05.069. Epub 2023 May 26. PMID 37267732
- [Derived] Vyas CM, Sadreyev RI, Gatchel JR, Kang JH, Reynolds CF, Mischoulon D, Chang G, Hazra A, Manson JE, Blacker D, De Vivo I, Okereke OI. Pilot Study of Second-Generation DNA Methylation Epigenetic Markers in Relation to Cognitive and Neuropsychiatric Symptoms in Older Adults. J Alzheimers Dis. 2023;93(4):1563-1575. doi: 10.3233/JAD-230093. PMID 37212116
- [Derived] Okereke OI, Vyas CM, Mischoulon D, Chang G, Cook NR, Weinberg A, Bubes V, Copeland T, Friedenberg G, Lee IM, Buring JE, Reynolds CF 3rd, Manson JE. Effect of Long-term Supplementation With Marine Omega-3 Fatty Acids vs Placebo on Risk of Depression or Clinically Relevant Depressive Symptoms and on Change in Mood Scores: A Randomized Clinical Trial. JAMA. 2021 Dec 21;326(23):2385-2394. doi: 10.1001/jama.2021.21187. PMID 34932079
- [Derived] Kang JH, Vyas CM, Okereke OI, Ogata S, Albert M, Lee IM, D'Agostino D, Buring JE, Cook NR, Grodstein F, Manson JE. Effect of vitamin D on cognitive decline: results from two ancillary studies of the VITAL randomized trial. Sci Rep. 2021 Dec 1;11(1):23253. doi: 10.1038/s41598-021-02485-8. PMID 34853363
- [Derived] Okereke OI, Reynolds CF 3rd, Mischoulon D, Chang G, Vyas CM, Cook NR, Weinberg A, Bubes V, Copeland T, Friedenberg G, Lee IM, Buring JE, Manson JE. Effect of Long-term Vitamin D3 Supplementation vs Placebo on Risk of Depression or Clinically Relevant Depressive Symptoms and on Change in Mood Scores: A Randomized Clinical Trial. JAMA. 2020 Aug 4;324(5):471-480. doi: 10.1001/jama.2020.10224. PMID 32749491
- [Derived] Donneyong M, Reynolds C, Mischoulon D, Chang G, Luttmann-Gibson H, Bubes V, Guilds M, Manson J, Okereke O. Protocol for studying racial/ethnic disparities in depression care using joint information from participant surveys and administrative claims databases: an observational cohort study. BMJ Open. 2020 Jan 7;10(1):e033173. doi: 10.1136/bmjopen-2019-033173. PMID 31915172
- [Derived] Okereke OI, Reynolds CF 3rd, Mischoulon D, Chang G, Cook NR, Copeland T, Friedenberg G, Buring JE, Manson JE. The VITamin D and OmegA-3 TriaL-Depression Endpoint Prevention (VITAL-DEP): Rationale and design of a large-scale ancillary study evaluating vitamin D and marine omega-3 fatty acid supplements for prevention of late-life depression. Contemp Clin Trials. 2018 May;68:133-145. doi: 10.1016/j.cct.2018.02.017. Epub 2018 Mar 8. PMID 29526608
- See also: Welcome to the VITAL study website — http://www.vitalstudy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 401605 initially screened; 39430 eligible to enter run-in; 25871 eligible for randomization; 2x2 factorial design: 12927 assigned to active vit D (of these, 6463 assigned to active omega-3 FAs and 6464 to placebo omega-3 FAs) & 12944 assigned to placebo vit D (of these, 6470 assigned to active omega-3 FAs and 6474 to placebo omega-3 FAs). Additional 7518 excluded per VITAL-DEP eligibility criteria; 18353 at risk for depression during follow-up.
Pre-assignment Details: The trial included a 3-month placebo run-in period to select participants likely to have adequate compliance. Only individuals who reported taking at least 2/3 of their study pills during the placebo run-in and met other eligibility criteria were randomized into the trial.
Groups:
- Vitamin D + Fish Oil Placebo: Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo
  vitamin D3: Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo: Fish oil placebo
- Vitamin D Placebo + Fish Oil: Vitamin D placebo
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  omega-3 fatty acids (fish oil): Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Vitamin D placebo: Vitamin D placebo
- Vitamin D Placebo + Fish Oil Placebo: Vitamin D placebo
  Fish oil placebo
  Fish oil placebo: Fish oil placebo
  Vitamin D placebo: Vitamin D placebo
- Vitamin D + Fish Oil: Vitamin D3 (cholecalciferol), 2000 IU per day
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  vitamin D3: Vitamin D3 (cholecalciferol), 2000 IU per day
  omega-3 fatty acids (fish oil): Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
Period: Overall Study
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil
Started | 4573 | 4563 | 4609 | 4608
Completed | 4573 | 4563 | 4609 | 4608
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil | Total
Number analyzed (Participants) | 4573 | 4563 | 4609 | 4608 | 18353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1642 | 1657 | 1674 | 1644 | 6617
  >=65 years | 2931 | 2906 | 2935 | 2964 | 11736
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.0) | 67.4 (7.1) | 67.5 (7.0) | 67.5 (7.1) | 67.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2261 | 2218 | 2265 | 2279 | 9023
  Male | 2312 | 2345 | 2344 | 2329 | 9330
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Total | 4573 | 4563 | 4609 | 4608 | 18353
  Non-Hispanic White | 3255 | 3266 | 3279 | 3297 | 13097
  Black or African-American | 855 | 833 | 869 | 850 | 3407
  Hispanic (not Black or African-American) | 185 | 170 | 176 | 177 | 708
  Asian or Pacific Islander | 66 | 72 | 78 | 78 | 294
  Native American or Alaskan Native | 37 | 39 | 33 | 41 | 150
  Other/Unknown | 175 | 183 | 174 | 165 | 697
Region of Enrollment [Number; unit: participants]
  United States | 4573 | 4563 | 4609 | 4608 | 18353

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Depression Event
Description: Depression syndrome will be determined by presence of clinical diagnosis, treatment and/or above-threshold symptoms on mood questionnaire (e.g., PHQ) items. This is an event outcome, where the depression event was defined as a new self-report of physician/clinician-diagnosed depression, treatment (medication and/or counseling) for depression, or presence of clinically relevant depressive symptoms (PHQ-8 total score >=10 points) on the annual study questionnaires that were administered over a median 5.3 years of randomized treatment and follow-up. Participants were followed for the depression event until the occurrence of the endpoint, death, or the end of the trial, whichever came first. The Outcome Measure table shows the counts of depression events in each randomized group by treatment.
Time Frame: From date of randomization until the date of the occurrence of the endpoint, death, or the end of the trial, whichever came first, assessed up to a median of 5.3 years of follow-up
Population: Analysis population reflects the randomized groups by treatment agents, as all published analyses per protocol were conducted comparing active treatment to placebo. These groups were: n=9181 randomized to active vitamin D and n=9172 randomized to vitamin D placebo; n=9171 randomized to active fish oil and n=9182 randomized to fish oil placebo. Per intervention results are presented for active vitamin D vs. matching vitamin D placebo and for active fish oil vs. matching fish oil placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin D: Vitamin D3: Vitamin D3 (cholecalciferol), one 2000 IU capsule per day
- Vitamin D Placebo: Vitamin D placebo: Vitamin D placebo, one capsule per day
- Active Fish Oil: Fish oil: Omacor, one capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
- Fish Oil Placebo: Fish oil placebo: Fish oil placebo, one capsule per day
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 9181 | 9172 | 9171 | 9182
Participants | 609 | 625 | 651 | 583
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p = 0.62, Regression, Cox — P-value was not adjusted for multiple comparisons. A priori, two-sided tests with an alpha level of 0.025 were used to account for the 2 co-primary outcomes (depression event and mood scores); Hazard Ratio (HR) = .97, 95% CI 2-sided [.87 to 1.09] — Active treatment vs. Placebo comparison
Statistical Analysis 2: Comparison: Active Fish Oil vs Fish Oil Placebo; Test type: Superiority; p = 0.03, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [1.01 to 1.26] — Active treatment vs. Placebo comparison

2. Primary Outcome: Mood Scores
Description: Mood scores are evaluated by the 8-item Patient Health Questionnaire (PHQ-8). The measured outcome was the total PHQ-8 score. The PHQ-8 includes items corresponding to the criteria for major depression. Each of the 8 items can be scored as 0, 1, 2, or 3 points (higher score means worse symptoms). The 8 items are summed to a total PHQ-8 score. The range for the PHQ-8 score is 0-24 points; higher scores denote worse mood or depressive symptoms. The PHQ-8 was measured annually at baseline and at up to 5 follow-up times (for a maximum of 6 time points). Data from all time points was used to determine the mean differences in change in mood scores over all follow-up by randomized treatment. Per protocol, the Statistical Analysis section shows the results for the primary outcome of mean difference in overall change in PHQ-8 scores comparing active and placebo groups (for each agent).
Time Frame: Baseline, follow-up year 1, follow-up year 2, follow-up year 3, follow-up year 4, and follow-up year 5
Population: Analysis population reflects the randomized groups by treatment agents, as all published analyses per protocol were conducted comparing active treatment to placebo. These were n=9181 randomized to active vitamin D; n=9172 randomized to vitamin D placebo; n=9171 randomized to active fish oil; n=9182 randomized to fish oil placebo. Per intervention results are presented for active treatment vs placebo. Each row shows exact number of participants providing responses to the PHQ-8 at that timepoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 9181 | 9172 | 9171 | 9182
score on a scale
  Baseline adjusted mean | 1.08 [1.05 to 1.11] | 1.13 [1.09 to 1.16] | 1.09 [1.06 to 1.13] | 1.11 [1.08 to 1.15]
  Mean change at Year 1: number analyzed (Participants) | 8534 | 8486 | 8471 | 8549
  Mean change at Year 1 | 0.03 [-0.01 to 0.07] | 0.03 [0.00 to 0.07] | 0.05 [0.01 to 0.09] | 0.01 [-0.02 to 0.05]
  Mean change at Year 2: number analyzed (Participants) | 8381 | 8344 | 8354 | 8371
  Mean change at Year 2 | 0.07 [0.03 to 0.11] | 0.04 [0.00 to 0.08] | 0.07 [0.03 to 0.11] | 0.04 [0.00 to 0.08]
  Mean change at Year 3: number analyzed (Participants) | 8176 | 8112 | 8116 | 8172
  Mean change at Year 3 | 0.09 [0.05 to 0.13] | 0.07 [0.03 to 0.12] | 0.10 [0.06 to 0.15] | 0.06 [0.02 to 0.10]
  Mean change at Year 4: number analyzed (Participants) | 7763 | 7603 | 7676 | 7690
  Mean change at Year 4 | 0.06 [0.02 to 0.10] | 0.07 [0.03 to 0.11] | 0.08 [0.04 to 0.12] | 0.05 [0.01 to 0.09]
  Mean change at Year 5: number analyzed (Participants) | 5316 | 5231 | 5295 | 5252
  Mean change at Year 5 | 0.20 [0.15 to 0.25] | 0.16 [0.11 to 0.22] | 0.18 [0.13 to 0.23] | 0.19 [0.13 to 0.24]
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test of whether the mean difference in change comparing the treatment groups is different than zero. See full SAP for all details; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.04 to 0.05]
Statistical Analysis 2: Comparison: Active Fish Oil vs Fish Oil Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.01 to 0.07]

3. Other Pre Specified Outcome: Number of Participants With an Incident Depression Event
Description: Post-hoc Outcome. Incident Depression is defined as depression cases that occurred among those with no past history of depression as of baseline. Incident depression event was determined by presence of clinical diagnosis, treatment and/or above-threshold symptoms on mood questionnaire (i.e., PHQ-8 >=10 points).
Time Frame: as for outcome 1
Population: Post-hoc Outcome. Incident Depression is defined as depression cases that occurred among those with no past history of depression as of baseline. Incident depression event was determined by presence of clinical diagnosis, treatment and/or above-threshold symptoms on mood questionnaire (i.e., PHQ-8 >=10 points). Among the n=18,353 participants randomized, there were n=16657 without a history of depression at baseline and therefore at risk for incident depression.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 8350 | 8307 | 8322 | 8335
Participants | 459 | 461 | 493 | 427
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; Test type: Superiority; p = 0.88, Regression, Cox — P-value not adjusted for multiple comparisons. This outcome was not a pre-specified primary outcome and results are to be interpreted with caution; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.87 to 1.13] — Active treatment vs. Placebo comparison
Statistical Analysis 2: Comparison: Active Fish Oil vs Fish Oil Placebo; Test type: Superiority; p = 0.02, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.03 to 1.33] — Active treatment vs. Placebo comparison

4. Other Pre Specified Outcome: Number of Participants With a Recurrent Depression Event
Description: Post-hoc Outcome. Recurrent depression is defined as depression cases that occurred among those with past history of depression, but not under treatment or active in the past 2 years as of baseline. Recurrent depression event will be determined by presence of clinical diagnosis, treatment and/or above-threshold symptoms on mood questionnaire (i.e., PHQ-8 >=10 points).
Time Frame: as for outcome 1
Population: Post-hoc Outcome. Recurrent Depression is defined as depression cases that occurred among those with past history of depression, but not active in the past 2 years as of baseline. Recurrent depression event will be determined by presence of clinical diagnosis, treatment and/or above-threshold symptoms on mood questionnaire (i.e., PHQ-8 >=10 points). Among n=18,353 randomized, n=1696 were eligible for recurrent depression.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 831 | 865 | 849 | 847
Participants | 150 | 164 | 158 | 156
Statistical Analysis 1: Comparison: Active Vitamin D vs Vitamin D Placebo; P-value not adjusted for multiple comparisons. This outcome was not a pre-specified primary outcome and results are to be interpreted with caution; Test type: Superiority; p = 0.67, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.76 to 1.19] — Active treatment vs. Placebo comparison
Statistical Analysis 2: Comparison: Active Fish Oil vs Fish Oil Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.88, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.82 to 1.27] — Active treatment vs. Placebo comparison

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire randomized treatment and follow-up period, which was a median of 5.3 years. VITAL-DEP is an ancillary study of the VITAL trial. For total adverse events reported by the parent VITAL trial, please see Results reported by VITAL, NCT01169259.
Description: Results for adverse events are reported by each of the 4 factorial arms of the trial.
Groups:
- Vitamin D + Fish Oil Placebo: Vitamin D: Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo: Fish oil placebo, one capsule per day
- Vitamin D Placebo + Fish Oil: Vitamin D placebo: Vitamin D3 placebo, one capsule per day
  Fish oil: Omacor, one capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
- Vitamin D Placebo + Fish Oil Placebo: Vitamin D placebo: Vitamin D3 placebo, one capsule per day
  Fish oil placebo: Fish oil placebo, one capsule per day
- Vitamin D + Fish Oil: Vitamin D: Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil: Omacor, one capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil
All-Cause Mortality (participants affected / at risk) | 153/4573 | 152/4563 | 133/4609 | 153/4608
Serious Adverse Events (participants affected / at risk) | 545/4573 | 569/4563 | 570/4609 | 549/4608
Other Adverse Events (participants affected / at risk) | 2803/4573 | 2789/4563 | 2876/4609 | 2825/4608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D + Fish Oil Placebo (N=4573) | Vitamin D Placebo + Fish Oil (N=4563) | Vitamin D Placebo + Fish Oil Placebo (N=4609) | Vitamin D + Fish Oil (N=4608)
Major cardiovascular event (Vascular disorders) | 144 | 129 | 126 | 120
Invasive cancer of any type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 281 | 301 | 291 | 312
Gastrointestinal Bleeding (Blood and lymphatic system disorders) | 111 | 133 | 135 | 107
Hypercalcemia (Endocrine disorders) | 47 | 49 | 53 | 42
Suicide (Psychiatric disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D + Fish Oil Placebo (N=4573) | Vitamin D Placebo + Fish Oil (N=4563) | Vitamin D Placebo + Fish Oil Placebo (N=4609) | Vitamin D + Fish Oil (N=4608)
Hyperparathyroidism or parathyroid condition (Endocrine disorders) | 19 | 17 | 27 | 10
Kidney stones (Renal and urinary disorders) | 172 | 131 | 163 | 158
Kidney failure (Renal and urinary disorders) | 27 | 28 | 29 | 19
Hematuria (Blood and lymphatic system disorders) | 319 | 293 | 318 | 333 — Blood in urine
Easy bruising (Blood and lymphatic system disorders) | 1167 | 1124 | 1141 | 1152
Frequent nosebleeds (Blood and lymphatic system disorders) | 159 | 158 | 163 | 159
Stomach upset or pain (Gastrointestinal disorders) | 1594 | 1616 | 1625 | 1615
Skin rash (Skin and subcutaneous tissue disorders) | 1105 | 1169 | 1184 | 1124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT01696435/Prot_SAP_000.pdf